CLINICAL TRIAL: NCT04184778
Title: Does Tracheal Tube Size Affect Patient's Experience of Postoperative Sore Throat and Hoarseness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Associate professor, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHN_DMK_06
Record Dates: First submitted 2019-04-10; First posted 2019-12-04 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Sore Throat; Hoarseness
Keywords: postoperative; Tube size; Patient experience
MeSH Terms: conditions — Pharyngitis; Hoarseness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Woman tube size 6.0 (Experimental): Smaller tube than normal
  Interventions: Device: Smaller tube size
- Woman tube size 7.0 (No Intervention): Usual tube size
- Man tube size 7.0 (Experimental): Smaller tube than normal
  Interventions: Device: Smaller tube size
- Man tube size 8.0 (No Intervention): Usual tube size

INTERVENTIONS:
Device: Smaller tube size — Comparing how tube size affect patient's experience of postoperative sore throat and hoarseness in men and women.
  Arms: Man tube size 7.0; Woman tube size 6.0

SUMMARY:
How tube size affect patient's experience of postoperative sore throat and hoarseness

DETAILED DESCRIPTION:
A randomised controlled study studying how tube size affect patient's experience of postoperative sore throat and hoarseness.

The patients are randomised on the basis of gender. Men are randomized to tube size 8.0 (usual) or 7.0. Women are randomized to tube size 7.0 (usual) or 6.0.

ELIGIBILITY:
Inclusion Criteria:

* Need for intubation
* Elective surgery
* ASA Group I and II
* Understands and speaks Danish
* give one's consent

Exclusion Criteria:

* Known dementia
* SARI score >4
* BMI > 35
* Acute intubation
* attempt intubation > 2
* known with previously difficult intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 261 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Sore throat after intubation | 7 days
  Survey - experienced postoperative sore throat after intubation. A scale from 1-4 is used; 1 indicated no sore throat and 4 indicated seriously sore throat.
Hoarseness after intubation | 7 days
  Survey - experienced postoperative hoarseness after intubation. A scale from 1-4 is used; 1 indicated no hoarseness and 4 indicated seriously hoarseness.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte M Kristensen, PhD, Principal Investigator — Regionshospital Nordjylland
Locations (2):
- Denmark (2):
  - North Denmark Regional Hospital, Hjørring
  - Aalborg University Hospital, Thisted